CLINICAL TRIAL: NCT06711029
Title: Effect of Different Duration and Number of Passive Ultrasonic Irrigation Activation Cycles on Postoperative Pain in Teeth with Symptomatic Irreversible Pulpitis: a Randomized Clinical Trial
Brief Title: Effect of Passive Ultrasonic Irrigation Activation Cycle on Postoperative Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esin Özlek (Other)
Collaborators: Yuzuncu Yil University (Other)
Responsible Party: Sponsor-Investigator, Esin Özlek, Associate professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03/15.11.2023
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Passive ultrasonic irrigation; Activation cycles
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 3 groups according to the final irrigation activation method; Group 1: Control Group, Group 2: Passive Ultrasonic Irrigation 3*20 sec, Group 3: Passive Ultrasonic Irrigation 6*10 sec.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Active Comparator): In the final irrigation, 6 ml of 5.252% NaOCI will be applied with needle irrigation for a total of 60 seconds.
  Interventions: Other: Conventional needle irrigation
- Passive Ultrasonic Irrigation 3*20 sec (Active Comparator): In the final irrigation, 6 ml of 5.25% NaOCI will be applied as 3*20 seconds with PUI for a total of 60 seconds.
  Interventions: Other: Passive Ultrasonic Irrigation with 3*20 sn
- Passive Ultrasonic Irrigation 6*10 sec (Active Comparator): In the final irrigation, 6 ml of 5.25% NaOCI will be applied as 6*10 seconds with PUI for a total of 60 seconds.
  Interventions: Other: Passive Ultrasonic Irrigation with 6*10 sn

INTERVENTIONS:
Other: Conventional needle irrigation — Conventional needle irrigation method was applied. As a final irrigation, 6 ml NaOCl was applied with 60 seconds of needle irrigation followed by 60 seconds of rest.
  Arms: Control Group
Other: Passive Ultrasonic Irrigation with 3*20 sn — In the final irrigation, 6 ml (3×2 ml) NaOCl was activated by PUI for 20 seconds in 3 cycles (60 seconds total). Before each cycle, 2 ml of NaOCl solution was refreshment.
  Arms: Passive Ultrasonic Irrigation 3*20 sec
Other: Passive Ultrasonic Irrigation with 6*10 sn — For the final irrigation, 6 ml (6×1 ml) NaOCl was activated with PUI for 10 seconds in 6 cycles (60 seconds total). Before each cycle, 1 ml of NaOCl solution was refreshment.
  Arms: Passive Ultrasonic Irrigation 6*10 sec

SUMMARY:
One of the most important goals of root canal treatment is to eliminate bacteria from infected canals. However, conventional irrigation methods combined with mechanical preparation applied during root canal treatment may not be sufficient for optimal disinfection. Various studies have shown that there are areas in the root canal that cannot be reached during chemomechanical shaping. One of the most popular techniques developed to deliver irrigation solutions to these areas is the Passive Ultrasonic Irrigation (PUI) technique, which provides good efficiency in terms of cleaning the root canal system. Activation of NAOCI with ultrasonic systems in the final irrigation significantly reduces the amount of microorganisms in the canal. Although the use of PUI in the final irrigation increases the effectiveness of irrigation solutions and enables the solutions to reach the apical third of the root canal, it causes extrusion of solutions into periapical tissues, albeit in small amounts, due to the positive apical pressure it creates during irrigation, and this causes postoperative pain. Postoperative pain is an undesirable but frequently encountered condition after endodontic treatment. During root canal treatment, extrusion of irrigation solutions or debris from the apex, mechanical, chemical or microbial factors can cause postoperative pain. In one study, the incidence of postoperative pain after endodontic treatment was reported to vary from 3% to 58%. Although the most effective is not yet fully known, when the literature is reviewed, different durations and cycles have been used for PUI. The change in the number of PUI cycles increases the microflow in the root canal, which may increase irrigation extrusion from the apical region and affect postoperative pain. Although many results have been reported in studies comparing the effect of final activation with Passive Ultrasonic Irrigation on postoperative pain with another technique, the activation cycle with PUI was determined as 3 times and 20 seconds each time, and this cycle order remained the same most of the time. Since there is no study in which the differences between cycles in activation with PUI affected postoperative pain, in this study the irrigation solution will be activated with PUI 3 times for 20 seconds and 6 times for 10 seconds, and the postoperative pain created by these two cycle orders will be compared.

DETAILED DESCRIPTION:
The study is planned to be conducted on 60 patients between the ages of 18-45 who were diagnosed and followed up at the Endodontics Clinic of the Faculty of Dentistry of Van Yuzuncu Yil University. Patients with no systemic disease, diagnosed with irreversible pulpitis, single-rooted and single-canal lower premolar teeth will be included in the case group. Patients with resorption and calcification at the roots of their teeth, incomplete root development, pregnant and breastfeeding, those who have taken analgesics or anti-inflammatory drugs in the last 12 hours, those who have used antibiotics in the last month, and those who cannot use a rubber dam in root canal treatment will not be included in the study. After obtaining the consent form from the patients, local anesthesia (Ultracain DS Fort, Hoechst-Marian Roussel, Frankfurt, Germany) will be applied to the tooth to be treated with root canal treatment. The access cavity will be opened with diamond burs under rubber dam isolation. The working length will be determined using a #10 K file (Mani Inc, Tochigi, Japan) and an electronic apex locator (Propex Pixi, Dentsply Maillefer, Switzerland). The root canals will be shaped to a size 40/0.06 using NiTI rotary files (ProTaper Next; Dentsply Sirona) at 300 rpm and 2 Ncm according to the manufacturer's instructions. The patients will be divided into 3 groups according to the final irrigation activation protocol for root canal treatment: Group 1: Control group. In the final irrigation, NaOCI will be applied with needle irrigation for a total of 60 s. Group 2: PUI 3*20 s. In the final irrigation, NaOCI will be applied with PUI for 3*20 s for a total of 60 s. Group 3: PUI 6*10 s. In the final irrigation, NaOCI will be applied for 60 seconds in total with PUI for 6*10 seconds. 5.25% NaOCI and 17% EDTA will be used as irrigation solution during the shaping process. NaviTip irrigation needle (30-G; Ultradent Products Inc, South Jordan, USA) will be used in the irrigation process during shaping. After the activation process is completed, the canals will be rinsed with distilled water as the final irrigation and the root canals will be filled with gutta percha and Adseal (Meta Biomed, Cheongju, North Korea) root canal sealer using the single cone method. The teeth will be restored with composite. Patients will be prescribed 400 mg ibuprofen anti-inflammatory medication to use in case of severe pain. The pain levels of the patients before and after the procedure will be evaluated with the VAS (Visual Analogue Scale) pain scale. Patients will be given a 10 cm paper ruler to record their pain levels at 6, 12, 24, 48, 72 hours and 1 week. Patients will be instructed on how to score their pain levels and will be asked to mark their pain levels on the ruler at the specified hours. At the end of the 1 week period, the rulers will be collected from the patients and the data will be statistically analyzed and interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 45 years
* Single-rooted and single-canal mandibular premolars diagnosed with symptomatic irreversible pulpitis

Exclusion Criteria:

* Patients who are taken analgesic inflammatory drugs with in the last 12 hours
* Pregnancy or lactation
* Teeth with calcified canals
* Teeth with sensitive to percussion and palpation
* Teeth with root resorption
* Teeth with immature/open apex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score Scala | The change in the postoperative pain levels by the patient at the 6 hours, 12 hours, 24 hours, 48 hours, 72 hours and at the end of 1 week will be compared.
  Postoperative pain will be assessed with a visual analog score after endodontic treatment. Scores will be given between 0-10. A score of '0' means no pain, a score of '10' means very severe pain. The higher the score, the higher the pain level.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Topcuoglu HS, Topcuoglu G, Arslan H. The Effect of Apical Positive and Negative Pressure Irrigation Methods on Postoperative Pain in Mandibular Molar Teeth with Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2018 Aug;44(8):1210-1215. doi: 10.1016/j.joen.2018.04.019. Epub 2018 Jun 20. PMID 29935873
- [Background] Estevez R, Conde AJ, Valencia de Pablo O, de la Torre F, Rossi-Fedele G, Cisneros R. Effect of Passive Ultrasonic Activation on Organic Tissue Dissolution from Simulated Grooves in Root Canals Using Sodium Hypochlorite with or without Surfactants and EDTA. J Endod. 2017 Jul;43(7):1161-1165. doi: 10.1016/j.joen.2017.01.041. Epub 2017 Apr 14. PMID 28416316
- [Background] Middha M, Sangwan P, Tewari S, Duhan J. Effect of continuous ultrasonic irrigation on postoperative pain in mandibular molars with nonvital pulps: a randomized clinical trial. Int Endod J. 2017 Jun;50(6):522-530. doi: 10.1111/iej.12666. Epub 2016 Jun 28. PMID 27248848
- [Background] Ali A, Hashem AAR, Roshdy NN, Abdelwahed A. The Effect of Final Irrigation Agitation Techniques on Postoperative Pain after Single Visit Root Canal Treatment of Symptomatic Irreversible Pulpitis: A Randomised Clinical Trial. Eur Endod J. 2023 May;8(3):187-193. doi: 10.14744/eej.2022.39200. PMID 37257031